CLINICAL TRIAL: NCT04966858
Title: Renewal of the Multi-center Randomized Controlled Trial of Refeeding in Anorexia Nervosa
Brief Title: Individualized Study of Refeeding to Optimize iNpatient Gains
Acronym: i-STRONG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01HD082166-06A1 (NIH); 20-32551 (Other: UCSF IRB); R01HD082166 (NIH); HD082166 (Other: Federal Identifier, per NIH application); P0547076 (Other: NIH Application Identifier)
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atypical Anorexia Nervosa
Keywords: Malnutrition; Refeeding; Nutritional Rehabilitation; Adolescent Medicine
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants will be recruited upon hospital admission at the University of California, San Francisco (UCSF) and Stanford and randomly assigned to Individualized Caloric Refeeding (ICR) or Higher Calorie Refeeding (HCR) for the duration of the hospitalization. Treatment ends at hospital discharge with open follow-up for one year. Participants followed daily in hospital and at 3mo, 6mo, 9mo, and 12mo post-discharge.
Masking Description: Treatments are not to be blinded, since both the patients and clinicians who work with this population are highly skilled at estimating kcal and would be able to determine group assignment by simply viewing meal trays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Caloric Refeeding (ICR) (Experimental): Starting 50 kcal/kg/d, increasing by 200 kcal/d to goal
  Interventions: Other: Individualized Caloric Refeeding (ICR)
- Higher Calorie Refeeding (HCR) (Active Comparator): Starting 2000 kcal/d, increasing by 200 kcal/d to goal
  Interventions: Other: Higher Calorie Refeeding (HCR)

INTERVENTIONS:
Other: Individualized Caloric Refeeding (ICR) — Meal-based refeeding in hospital, starting at 50 calories per kilogram of body weight, and increasing by 200 calories per day until caloric goal achieved
  Other Names: ICR
  Arms: Individualized Caloric Refeeding (ICR)
Other: Higher Calorie Refeeding (HCR) — Meal-based refeeding in hospital, starting at 2000 calories per day, and increasing by 200 calories per day until caloric goal achieved
  Other Names: HCR
  Arms: Higher Calorie Refeeding (HCR)

SUMMARY:
The primary purpose of the trial is to compare the efficacy and safety of Individualized Caloric Refeeding (ICR) to the new standard of care, Higher Calorie Refeeding (HCR), in hospitalized patients with atypical anorexia nervosa (AAN), and clinical remission over one year of follow-up.

DETAILED DESCRIPTION:
Atypical Anorexia Nervosa (AAN) is a new diagnosis describing patients with malnutrition and significant weight loss yet "normal" weight. These patients responded poorly to HCR, the superior refeeding treatment in the parent trial, which was designed for low-weight patients with typical AN. The proposed trial will examine the safety and efficacy of a new treatment for AAN with the potential to improve treatment outcomes for this diverse and growing patient population. The major finding motivating the proposed trial is that participants with AAN gained weight 40 percent slower and required 3.0 additional days in hospital to restore medical stability on HCR, as compared to AN. The research team has developed Individualized Caloric Refeeding (ICR), which doses calories to weight consistent with other pediatric treatments (e.g. medication).

The primary purpose of the proposed trial is to compare the efficacy and safety of ICR to the new standard of care (HCR) in hospitalized patients with AAN. The investigators hypothesize that ICR will restore medical stability faster than HCR with no increase in electrolyte abnormalities. After hospitalization, the major barrier to care in AAN is lack of consensus on clinical remission and whether these formerly overweight patients should gain weight to recover. The research team will examine metabolic, hormonal and psychological markers during long-term follow-up, toward the goal of developing a definition of clinical remission in AAN.

Design Summary: Randomized controlled trial in N=74 participants age 12-24 with AAN, consented upon hospital admission, randomly assigned to ICR or HCR, followed daily in hospital and at 3, 6, 9 and 12 mo.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-24 yrs
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for AAN
* Hospitalized with medical instability, as defined by:

  1. night time heart rate (HR) <45 bpm,
  2. systolic blood pressure (SBP) <90 mmHg,
  3. temperature <35.6° C,
  4. orthostatic Δ HR >35 bpm, or
  5. orthostatic Δ SBP >20 mmHg

Exclusion Criteria:

* Bulimia nervosa
* Current pregnancy
* Chronic disease (e.g. immune, renal disease)
* Acute/active suicidality or psychosis
* Hospital admissions for refeeding in the prior 6 mo.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to Achieve Medical Stability in Hospital | Inpatient hospitalization from day of admission to day of discharge, average 1-2 weeks
  Medical stability will be adjudicated by a five-point index: (1) 24 hour heart rate of 45 beats/min or more, (2) systolic blood pressure of 90 millimeters of mercury (mmHg) or more, (3) temperature of 35.6° C or more, (4) orthostatic increase in heart rate of 35 beats/min or less, (5) orthostatic change in systolic blood pressure of 20 mmHg or less.

SECONDARY OUTCOMES:
Incidence of low serum electrolytes during refeeding in hospital | Inpatient hospitalization from day of admission to day of discharge, average 1-2 weeks
  Incidence of low electrolytes will be defined as: (1) hypophosphatemia less than 3 milligrams per deciliter (mg/dL), (2) hypomagnesaemia less than 1.8 mg/dL, and (3) hypokalemia less than 3.5 milliequivalent per liter (mEq/L) during hospitalization.

OTHER OUTCOMES:
Percentage median BMI (mBMI) Over 12 Months | 12 months post-study hospitalization
  Measured BMI will be divided by the mBMI for age and sex per national growth data to give the percentage mBMI.
Eating Disorder Examination Questionnaire (EDE-Q) Score Over 12 Months | 12 months post-study hospitalization
  The EDE-Q will be self-administered; scores range from 1 to 6, with higher scores indicating greater severity and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K Garber, RD, PhD, Principal Investigator — University of California, San Francisco; Neville H Golden, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Lucille Packard Children's Hospital, Palo Alto, California
  - University of California, San Francisco Benioff Children's Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: No